CLINICAL TRIAL: NCT00343993
Title: Noninvasive Positive Pressure Ventilation for ALI/ARDS:a Multicentre Randomized Controlled Trial
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y0905001040291
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Last update posted 2007-04-04 (Estimated); Status verified 2007-04

CONDITIONS: Acute Lung Injury; Acute Respiratory Distress Syndrome
Keywords: noninvasive positive pressure ventilation; acute lung injury; acute respiratory distress syndrome
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: noninvasive positive pressure ventilation

SUMMARY:
with appropriate inspired oxygen concentrations, NPPV would prevent intubation and hence avert the poor outcome associated with the need of invasive ventilation in patients with ALI/ARDS.

DETAILED DESCRIPTION:
Noninvasive positive-pressure ventilation (NPPV) is increasingly being used in the care of patients suffering acute respiratory failure. High-level evidence supports the use of NPPV to treat exacerbation of chronic obstructive pulmonary disease (COPD). More recently, NIV has shown to reduce the need for intubation in selected groups of patients with severe cardiogenic pulmonary edema, immunosuppression, and respiratory failure after lung resection. In their subgroup analysis of the five randomized control trials, however, patients with acute lung injury (ALI) or ARDS still couldn't avoid intubation and death even treated with NPPV. Till now, there has been no randomized controlled study of NPPV in patients with ALI or ARDS. We hypothesized that in patients with ALI/ARDS, early use of NPPV, providing appropriate inspired oxygen concentrations, would prevent intubation as the primary end-point variable, hence avert the poor outcome associated with the need of invasive ventilation. Accordingly, we conducted a prospective, randomized controlled trial to assess the efficacy of NPPV compared with a standard regime consisting of high-concentration oxygen therapy.

ELIGIBILITY:
Inclusion Criteria:

* Meet the ALI/ARDS criteria

Exclusion Criteria:

* Age > 85
* pH < 7.35 or PaCO2 >50mmHg
* Glasgow Coma Scale (GCS)<11
* Airway or facial deformity
* Pneumothorax or pneumomediastinum
* Unable to spontaneously clear secretions from their airway
* Respiratory arrest
* Shock or hemodynamic instability (systolic blood pressure <90 mmHg associated with decreased urinary output (<20 mL.h-1) despite fluid repletion and use of vasoactive agents) of other causes
* Severe ventricular arrhythmia or active myocardial ischemia
* Severe organ dysfunction (including gastrointestinal hemorrhage, disseminated intravascular coagulation, hepatic and renal dysfunction, SOFA score>1)
* End-stage patients who are expected to survive less than six months
* Severe abdominal distension
* Refuse to receive NPPV
* Unable to cooperate with the application of NPPV

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2006-06; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
The intubation rate who meet the intubation criteria predefined

SECONDARY OUTCOMES:
Mortality in the ICU and hospital

CONTACTS AND LOCATIONS:
Overall Officials: Wang Chen, MD, Study Chair — Beijing Chao Yang Hospital
Locations (1):
- Beijing chaoyang hospital-affiliate of capital medical university, Beijing, China